CLINICAL TRIAL: NCT01281891
Title: Postoperative Pain Relief Following Total Hip Arthroplasty. A Comparison Between Intrathecal Morphine (IM) and Local Infiltration Analgesia (LIA)
Acronym: HÖFTPLASTIK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Per Essving, Assistant Professor, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THA001
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Primary Osteoarthritis Requiring Total Hip Replacement
Keywords: Drug: Morphine intrathecal; Pain: Postoperative; Surgery: Total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local Infiltration Analgesia (Experimental): Combination of ropivacaine, ketorolac and adrenaline
  Interventions: Drug: LIA
- Intrathecal morphine (Active Comparator): Morphine special (preservative-free) injected intrathecally
  Interventions: Drug: I/T morphine

INTERVENTIONS:
Drug: LIA — Ropivacaine 0.2% Ketorolac 30 mg Adrenaline 0.1 mg/ml
  Arms: Local Infiltration Analgesia
Drug: I/T morphine — Morphine special 0.1 mg injected intrathecally
  Arms: Intrathecal morphine

SUMMARY:
Postoperative pain following total hip arthroplasty (THA) (1) is often considered moderate to severe and can therefore influence the postoperative course of event and result in delayed postoperative mobilization and prolonged hospitalization. It is therefore necessary to find the most optimal method for alleviation of pain for these patients. Traditionally, this has been managed by epidural analgesia, continuous peripheral nerve blocks, parental- or spinal opioids. Recently, Drs Kerr and Kohan at the Joint Orthopaedic Centre in Sydney, Australia developed a local infiltration analgesia (LIA) technique. The technique was introduced in Scandinavia during 2001 and has been shown to be efficacious during knee surgery. The LIA technique is based on a systemic infiltration of a mixture of a long-acting local anaesthetic (ropivacaine), a non steroidal anti-inflammatory drug (ketorolac), and epinephrine into the tissue around the surgical field to achieve satisfactory pain control with little physiological disturbance. A catheter is left from the skin and into the joint cavity, allowing repeated injection on the morning after surgery (10). Effective pain relief with early mobilization and reduced hospital stay has been reported following total knee arthroplasty and, recently, following unicompartmental knee arthroplasty.

The aim of this study is to assess whether LIA technique is equi-efficacious to intrathecal morphine, the standard of care in our hospital.

DETAILED DESCRIPTION:
This is a randomized, double blind parallel-group study where two different methods for postoperative pain relief after total hip arthroplasty, intrathecal morphine (IM) and local infiltration analgesia (LIA), will be assessed.

The study will be conducted at the Department of Anaesthesiology and Intensive Care and the Department of Orthopaedic Surgery, at USÖ. A total of 80 patients undergoing total hip arthroplasty will be included in the study, 40 patients in group IM and 40 patients in group LIA. The patients will be divided into one of the two groups according to computer-generated randomization. Study duration per patient will be 6 months.

Screening on the basis of inclusion and exclusion criteria will take place at the preoperative assessment at the outpatients' anesthesia clinic 3 - 6 weeks before the total hip arthroplasty. One of the participating investigators will inform the patient, both verbally and in writing, about what participation in the study involves. The patient will be given time to ask questions and to consider participation in the study.

If the patient wants to be enrolled in the study, inclusion will take place at the preoperative assessment that takes place before the total hip arthroplasty. One of the participating Investigators would inform the patient again about what participation in the study means. The patient will be given time to ask questions and to consider participation in the study. The patient can be enrolled in the study after signing and dating the written Informed Preoperative Preparation The patients will be informed in details about the surgery, anesthesia, postoperative pain relief and physiotherapy. All patients will be asked to complete two health related quality of life questionnaires, SF-36 and EQ5D (appendix 2 and 3).

A baseline value for HOOS (appendix 4) and NRS (Numeric Rating Score) will be assessed prior to surgery. The patients will also be instructed on how to use the patient controlled analgesia (PCA) morphine pump that will serve as post-operative rescue medication in case of pain > 3 on the numeric rating scale (NRS) Dalteparin 5000 IU is administered subcutaneously once each evening for 10 days, starting the night before surgery for thrombo-prophylaxis.

Randomisation Randomisation will be made at the USÖ Hospital Pharmacy the day before surgery. The patients will be randomized into two groups, 40 patients in Group IM and 40 patients in Group LIA, according to computer-generated randomization.

The study medication/saline will be prepared, blinded and labeled by a pharmacist at the USÖ Hospital Pharmacy. The hospital pharmacy will send the double-blinded study medication/saline to the operating theater on the day of surgery. This way, double blinding will be ensured such that neither the patient nor the anaesthesiologists, the staff attending the surgery, the staff concerned with the postoperative care of the patients or the physiotherapist are aware of the group to which the patient has been randomized. The study medication/saline will be stored in room temperature in the operating theatre and will be given within one hour from the time it is received. Study medication/saline for the peri-articular injection on postoperative day one will be kept in a refrigerator at the Department of Anesthesiology and intensive care until it is to be given.

Anaesthesia All patients will receive a mixture of midazolam 0.03 mg/kg orally 1 hour before planned surgery. Cloxacillin 1g will be given intravenously before surgery and at 8, 16 and 24 h postoperatively. The operation will be performed using spinal anaesthesia, performed in the sitting position, using a 27G spinal needle. All patients will receive bupivacaine plain 5 mg/ml (17.5 mg = 3.5 ml) injected intrathecally. In addition, patients randomized to Group IM will receive morphine special 0.4 mg/ml (0.1 mg =0.25 ml) and patients randomized to Group LIA will receive an equivalent amount (= 0.25 ml) of normal saline. Total volume of injectate will for each patient be 3.75 ml.

Surgery and Perioperative Management The surgery will be performed in a standardized way according to routine at Örebro University hospital. At the end of surgery, and after the hip prosthesis is in place, patients in Group LIA would receive a total volume of 151.5 ml of a mixture consisting of: a long-acting local anaesthetic (ropivacaine 2 mg/ml = 150 ml), a no-steroidal anti-inflammatory drug (ketorolac 30 mg/ml = 1 ml), and epinephrine (1 mg/ml = 0.5 ml) injected intraarticularly and into the surrounding peri-articular tissues in a standardized way. Patients in Group IM would receive a similar volume (151.5 ml) of normal saline injected in the same way at similar sites in order to ensure double-blinding of all personnel involved in the study.

A multi-holed catheter (a peri-articular catheter) would be inserted into the tissue planes under direct vision in a standardized way before closing the wound and would be connected to a bacterial filter under sterile conditions. After the surgery the patient would be transferred to the post-anaesthesia care unit (PACU) and thereafter to the orthopaedic ward for further management.

During the first post-operative day, 24 hours after surgery the following solutions will be injected peri-articularly via the multi-holed catheter by a nurse who is blinded to the injectate:

Group LIA:

20 ml of ropivacaine (7.5 mg/ml)

1 ml ketorolac (30 mg/ml)

1 ml of epinephrine (0.1 mg/ml)

Group IM:

22 ml saline

Total volume of injectate will for each patient be 22 ml.

The multi-holed catheter would then be removed and the tip of the catheter sent for culture and sensitivity testing. Any evidence of fever or local or systemic infection will be recorded.

Pain Management All patients will receive 1 g paracetamol orally 4 times a day, starting on the morning of the operation.

A patient controlled analgesia (PCA) morphine pump (1 mg bolus dose, 6 min lock-out time) would be connected IV in all patients, and will serve as rescue medication in case of pain > 3 on the numeric rating scale (NRS; 0 = no pain, 10 = worst imaginable pain). The patients will be instructed on its use the day before surgery. If pain is < 4 during a 12 h period, the PCA-pump will be discontinued and tramadol 50 mg given orally up to 4 times/day as necessary as rescue medication for pain management. All patients would receive Paracetamol 1 g six-hourly as basal analgesic.

Mobilization and Home discharge The first attempt to mobilization will be made about 30 min after the peri-articularly injection of study medication/saline, 24 h after surgery. The patient will be asked to stand up and to walk 10 steps. If unsuccessful, another attempt will be made to mobilize the patient every 12 h until the patient can walk 10 steps. If the 12 h period is after 9 pm, the next attempt would be made on the following morning. Subsequently, mobilization will also be quantified using a TUG test (appendix 5) from postoperative day 1 until discharge

The patient will be discharged when the discharge criteria are fulfilled:

* Mild pain (NRS < 3) sufficiently controlled by oral analgesics
* Ability to walk with elbow crutches
* Ability to eat and drink without nausea or vomiting
* No signs of any surgical complications

The patient will also be asked to register pain (NRS) and analgesic consumption during the first 14 postoperative days and at week 2, 3 and 4. (appendix 6)

Recordings and Assessments (Flowchart, appendix 7)

Demographic data:

Age, gender, height and weight.

Length of stay at the hospital (LOS):

The number of postoperative days to home discharge, day 0 = the day of surgery would be recorded.

Home discharge criteria are:

* Mild pain (NRS < 3) sufficiently controlled by oral analgesics,
* Ability to walk with elbow crutches
* The patient can eat and drink without nausea or vomiting
* No signs of any surgical complications.

Pain:

Pain assessment will be recorded by NRS scale preoperatively and at 1, 4, 8, 12, 24, 36 and 48 hours postoperative, subsequently every 24 hour until the patient is discharged from hospital, on day 14 and 3 and 6 months postoperatively.

Pain will be assessed both at rest and on motion (after walking 10 steps).

Analgesic consumption:

Morphine consumption will be recorded during 0 - 4, 4 - 24 and 24-48 hours postoperatively.

Oral analgesic consumption will be recorded each day until home discharge. The patients will be asked to record their pain and analgesic consumption once each day for 14 days and weekly on weeks 2, 3 and 4.

Surgical outcomes:

The research nurse or physiotherapist will record the hip extension and flexion every 24 h until discharge and after 14 days, 3 and 6 months postoperatively.

TUG test will be performed från postoperative day 1 until discharge Patient satisfaction during the first 24 postoperative hours and after 7 days will be rated according to a satisfaction score: 1= poor, 2= satisfactory, 3= good and 4= excellent.

HOOS will be collected preoperatively, and at 2 weeks, 3 and 6 months postoperatively.

Health-related questionnaires:

The SF-36 and EuroQol (EQ-5D) questionnaires will be collected preoperatively and postoperatively on day 7 (only EQ-5D), 3 and 6 months.

The SF-36 is a validated health survey consisting of 36 questions that measure 8 health concepts: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations secondary to emotional problems (RE) and mental health (MH). Additionally, 2 summary scores are available: a standardized physical component (PCS) and a standardized mental component (MCS).

The EuroQol (EQ-5D) is a standardised instrument for use as a measure of health outcome. It provides a single index value from 0 to 1 where 0 represents death and 1 represents perfects health.

ELIGIBILITY:
Inclusion Criteria:

1. 60 - 80 year-old undergoing total hip arthroplasty.
2. ASA I - II (appendix 1).
3. Have signed and dated Informed Consent.
4. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Re-operation of a previous total hip arthroplasty.
2. Allergy/intolerance to local anaesthetics, Morphine, Adrenaline, Ketorolac or Ropivacaine.
3. Serious liver- or renal disease judged by the investigator to be of such dignity as to prevent inclusion into the study.
4. Serious heart disease judged by the investigator to be of such dignity as to prevent inclusion into the study,
5. Patients with chronic pain who are taking opiate analgesics regularly.
6. Major bleeding disorders
7. Chronic obstructive pulmonary disease (COPD)
8. Severe asthma that is difficult to treat
9. Limited breathing capacity due to muscular dystrophy
10. Sleep apnoea syndrome
11. Other contraindication to spinal anaesthesia such as spinal stenosis, local infection or contraindications to local anaesthetics.
12. Participation in another clinical medicinal trial during the last 30 days or where follow-up is not completed.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption postoperatively | During 0 -24 hours postoperatively
  Other than total morphine consumption, even pain intensity on movement would be considered to be an important parallel end-point.

SECONDARY OUTCOMES:
Pain intensity (NRS, Numeric Rating Score; 0-10) | 0 - 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University Hospital, Örebro, Sweden